CLINICAL TRIAL: NCT04808583
Title: Efficacy of At-origin Uterine Artery Ligation Compared to Conventional Post-cornual Pedicle Ligation in Reducing Operative Time During Total Laparoscopic Hysterectomy
Brief Title: Uterine Artery Ligation at Origin in Total Laparscopic Hystrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasser Elrefaey, Assistant Lecturer of obstetrics and gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UALO20
Record Dates: First submitted 2021-02-22; First posted 2021-03-22 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Uterine Diseases
Keywords: laparscopic hystrectomy uterine artery operative time
MeSH Terms: conditions — Uterine Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Active Comparator): conventional TLH with uterine artery ligation after the cornual pedicles
  Interventions: Procedure: conventional TLH with uterine artery ligation after the cornual pedicles
- Group (B) (Experimental): TLH with uterine artery ligation at its origin at the beginning of the operation
  Interventions: Procedure: TLH with uterine artery ligation at its origin at the beginning of the operation

INTERVENTIONS:
Procedure: TLH with uterine artery ligation at its origin at the beginning of the operation — After insertion of the ports and surveying the abdomen as in the conventional method a window will be created in the broad ligament to enter the retroperitoneal space with exposure of the iliac vessel and identification of the internal iliac artery and its anterior branch which give rise to the uterine artery. Blunt dissection continues with identification of the paravesical and the pararectal spaces. The ureter is identified medially and the uterine artery laterally and dissection of the ureter away from the uterine artery will be done, followed by sealing the uterine artery 2 mm from its origin from the anterior branch of internal iliac artery
  Arms: Group (B)
Procedure: conventional TLH with uterine artery ligation after the cornual pedicles — Coagulation and section of round ligaments will be performed about 2 to 3 cm from the pelvic wall using blunt tip laparoscopic sealer LigaSure COVIDIEN (5mm-37cm) with average of sealing cycle of 2 to 4 seconds and 40 watts , followed by opening the anterior leaflet of the broad ligament to the vesico-uterine peritoneal reflection, coagulation and section of the infundibulo-pelvic ligament (total hysterectomy with bilateral adnexectomy) or of the uteroovarian ligament and the fallopian tubes (total hysterectomy). Then opening the posterior leaflet of the broad ligament to the cervix, opening of the vesico-vaginal space and dissecting the bladder downwards will be done (Poojari et al., 2014).
  Coagulation and section of the uterine pedicles: performed on the ascending segment of the uterine artery, will be carried out in a progressive manner on both sides.
  Arms: Group (A)

SUMMARY:
The aim of the current study is to compare between the uterine artery ligation at its origin at the beginning of the operation and the conventional method after cornual pedicle regarding their efficacy to minimize operative time in patients undergoing total laparoscopic hysterectomy.

DETAILED DESCRIPTION:
1. Approval of the study protocol will be sought from ASUMH ethical committee.
2. The patients will be enrolled from the outpatient gynecology clinic of ASUMH.
3. History, examination and routine investigations will be done to identify eligible patients.
4. Written informed consent will be sought from the patients after proper counseling.
5. Randomization: It will be a quasi-randomized clinical trial.
6. Allocation: through "Alternation" method. Eligible patients will be randomized into one of the two study groups, where odd numbered patients (ex: patient number 1, 3, 5, etc. …) will be allocated to group (A) and even numbered patients (ex: patient number 2, 4, 6, etc. …) will be allocated to group (B) till full-filing the sample size. Before the operation, the patient will be allocated according to her number.
7. Blinding: the patient will not be aware of the method used (either the conventional method or the At-origin ligation method) (single blinded).
8. Patients who are randomized to group A will undergo TLH in the conventional method as follows:

   Positioning:The patient will be positioned in dorsal decubitus, under general anesthesia, with oral tracheal intubation. The legs will be positioned in 30°flexion; the arms along the body, and the buttocks extending slightly over the edge of the surgical table. The bladder will be catheterized. The surgeon will be positioned to the left of the patient, the primary assistant on the right, and the second assistant is responsible for uterine manipulation.

   Uterine Cannulation: Uterine cannulation will be performed using uterine manipulator. Hysterometry will be performed, the cervix will be dilated using Hegar dilators if needed, and the manipulator will be inserted under direct vision into the cervix.

   A Veress needle will be inserted at the umbilicus or supraumbilical site depending on the size of the uterus and abdomen will be insufflated with carbon dioxide at initial pressure of 20 mm Hg and maintenance at 15 mm Hg. A 10 mm trocar will be inserted blindly, and 10 mm telescope will be introduced through this port. Uterus and the adnexa will be visualized. Three additional 5mm ports are introduced: one along the left spino-umbilical line at the junction of medial 2/3rd and lateral 1/3rd, second port at right angles to the previous port, and a third 5 mm port placed around 2 cm below and to the right of umbilicus. The entire abdomen is surveyed before starting the procedure. The size of the uterus, presence of myomas, and adnexa and course of ureters are visualized (Poojari et al., 2014).

   Coagulation and section of round ligaments will be performed about 2 to 3 cm from the pelvic wall using blunt tip laparoscopic sealer LigaSure COVIDIEN (5mm-37cm) with average of sealing cycle of 2 to 4 seconds and 40 watts , followed by opening the anterior leaflet of the broad ligament to the vesico-uterine peritoneal reflection, coagulation and section of the infundibulo-pelvic ligament (total hysterectomy with bilateral adnexectomy) or of the uteroovarian ligament and the fallopian tubes (total hysterectomy). Then opening the posterior leaflet of the broad ligament to the cervix, opening of the vesico-vaginal space and dissecting the bladder downwards will be done (Poojari et al., 2014).

   Coagulation and section of the uterine pedicles: performed on the ascending segment of the uterine artery, will be carried out in a progressive manner on both sides.

   Vault will be cut laparoscopically using monopolar hook and the specimen will be detached completely. The uterus with cervix will be delivered vaginally. The vaginal vault will then be sutured with number 0 delayed absorbable suture (vicryl).
9. While patients randomized to group B will undergo TLH as follows:

   After insertion of the ports and surveying the abdomen as in the conventional method a window will be created in the broad ligament to enter the retroperitoneal space with exposure of the iliac vessel and identification of the internal iliac artery and its anterior branch which give rise to the uterine artery. Blunt dissection continues with identification of the paravesical and the pararectal spaces. The ureter is identified medially and the uterine artery laterally and dissection of the ureter away from the uterine artery will be done, followed by sealing the uterine artery 2 mm from its origin from the anterior branch of internal iliac artery. Dissecting the utero-vesical fold and pushing the bladder down will move the ureters laterally and decrease the risk of injuring them. The vasculature of the uterus will thus be secured, and this will be evidenced by the color change in the fundus, which will become pale. The cornual pedicles on one side (including the round ligament and either the utero-ovarian or infundibulopelvic ligments ) will then be desiccated and cut using the ligasure. The coagulated uterine pedicles will be cut. The utero-sacral and cardinal ligaments will be desiccated and cut. Then the opposite side pedicles will be taken care of. (Poojari et al., 2014).
10. The operative time will be calculated and the total blood loss will be measured from the suction apparatus keeping in mind the amount of fluid used during irrigation. The urinary catheter will be removed after 6 hours and liquid diet will be started after peristalsis is established as evidenced by audible intestinal sounds. Follow up vital data and postoperative pain by visual analogue score and measuring postoperative hemoglobin, the patient will be discharged the following day and called for follow-up after 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age group (35-70 years old).
2. Women consenting to have a total laparoscopic hysterectomy.

Exclusion Criteria:

1. Patients with relative contraindication to general anesthesia (e.g. chronic liver cell failure)(All laparoscopic procedures are done under GA).
2. Patients with contraindication to laparoscopic surgery (e.g. severe cardio-pulmonary dysfunction).
3. Bleeding tendency (e.g. anticoagulants, platelets disorders)(will affect the blood loss measurement)
4. Body mass index more than 35 Kg/m2(not suitable for laparoscopic surgeries as obesity affects airway pressure )
5. Uncorrected anemic patients (Hemoglobin < 10 gm. /dl).(will affect the outcomes eg :

Blood transfusion , hospital stay … etc )

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Operative time in minutes | Intraoperative (once for each patient starting from port insertion till disconnecting the uterus from the vagina .)
  starting from port insertion till disconnecting the uterus from the vagina

SECONDARY OUTCOMES:
Blood loss in millimeters | Intraoperative (once for each patient at the end of the operation .)
  blood loss in the operation will be measured from the suction apparatus keeping in mind the amount of fluid used during irrigation.
postoperative pain measured using visual analogue score. | 6 hours postoperative - 12 hours postoperative
  VAS : visual analogue score where (0): no hurt - (10) : Hurts worst
Hospital stay (in days) | "through study completion, an average of 1 year".
  hospital stay in days after the procedure .
Complications | during the procedure,immediately after the procedure .
  (visceral , bladder or ureteric injuries).

CONTACTS AND LOCATIONS:
Overall Officials: Hazem M Sammour, MD, Study Chair — Professor of Obstetrics and Gynecology
Locations (1):
- Ain shams maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No